CLINICAL TRIAL: NCT06058429
Title: Immunogenicity After Primary Immunization and Booster Immunization of Sabin Strain Inactivated Polio Vaccine (Vero Cells) in Infants and Young Children and Enterovirus Serological Monitoring Study
Brief Title: Immunogenicity of After Primary Immunization and Booster Immunization of sIPV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Jiangxi Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRO-sIPV-MA4001-1-JX
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Polio
Keywords: immunogenicity of sIPV; primary immunization; booster immunization; simulteneous immunization; serology of antibodies against enterovirus
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2-3 months infants group: Subjects in this group had recieved three dose of sIPV as primay immunization, and about half of them recieved DTaP simultaneously.
  Interventions: Other: no intervention
- 18 months children group: Subjects in this group had recieved one dose of sIPV as booster immunization, and about half of them recieved MMR or hepatitis A vacine(live-attenuated or inactivated) simultaneously.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study after vaccination, no intervention will be used

SUMMARY:
This study was conducted on the basis of "Safety Observation of Sabin Strain Inactivated Polio Vaccine (Vero Cell) on primary Immunization, Booster Immunization and Simultaneous Vaccination with Other Vaccines in Infants and Young Children(ID: PRO-sIPV-MA4001-JX). Blood samples were collected in about 200 qualified subjects 1-9 months after their last vaccination of sIPV. And immunogenicity of sIPV and other vaccines simultaneously administrated will be tested, the antibodies against enterovirus (including EV71、CA16、CA6 and CA10) will also be tested.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the previous study (ID: PRO-sIPV-MA4001-JX)
* Subjects in the Primay immunization group(aged 2-3 months) need to complete 3 doses of sIPV vaccination, and the simultaneous vaccination group DTaP needs to complete 3 doses of vaccination; the booster immunity group(aged more than 18 months) needs to complete sIPV vaccination, and the simultaneous vaccination group needs to complete the corresponding vaccination;
* There should be an interval of 1-9 months between the last dose of vaccination and the date of blood sample collection;
* The guardian of subjects need to agree to sign the informed consent form.

Exclusion Criteria:

* The interval between vaccination and blood collection is less than 1 month, or more than 9 months;
* Subjects were participating in other clinical studies of vaccines or drugs;
* Other conditions that make subjects unsuitable for participating in this study judged by investigator's

Ages: 2 Months to 27 Months | Sex: All
Age Groups: Child
Study Population: Subjects in the Primay immunization group(aged 2-3 months) need to complete 3 doses of sIPV vaccination, and the simultaneous vaccination group DTaP needs to complete 3 doses of vaccination; the booster immunity group(aged more than 18 months) needs to complete sIPV vaccination, and the simultaneous vaccination group needs to complete the corresponding vaccination
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Antibody positivity rate of sIPV vaccine after primary immunization in infants | 1 month
Antibody positivity rate of sIPV after booster immunization with sIPV vaccine in young children | 1 month
seropositive rate of antibodies against different enteroviruses (EV71/CA16/CA6/CA10) in infants and young children | 1 month

SECONDARY OUTCOMES:
GMT of sIPV vaccine after primary immunization in infants | 1 month
GMT of sIPV after booster immunization with sIPV vaccine in young children | 1 month
GMT of antibodies against different enteroviruses | 1 month

OTHER OUTCOMES:
Antibody positivity rate and GMC for pertussis, diphtheria and tetanus after full vaccination with DTaP vaccine in infants | 1 month
Antibody positivity rate and GMC of hepatitis A vaccine after full vaccination in young children | 1 month
Antibody positivity rate and GMT for measles, rubella, and mumps after full vaccination of MMR vaccine in young children | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Center for Disease Control and Prevention, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo S, Li Z, Zheng M, Wu F, Sun J, Tuo L, Li S, Li X, Wei L, Xia Z, Xie P, Chen X, Zhao Y, Gao Y, Yu D. Safety and 6-month immune persistence of inactivated poliovirus vaccine (Sabin strains) simultaneously administrated with other vaccines for primary and booster immunization in Jiangxi Province, China. Vaccine. 2024 Aug 30;42(21):126183. doi: 10.1016/j.vaccine.2024.126183. Epub 2024 Jul 31. PMID 39088987